CLINICAL TRIAL: NCT01237106
Title: In Vitro Maturation for Polycystic Ovary Syndrome (PCOS)- A Pilot Study
Brief Title: In Vitro Maturation (IVM) for Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Reproductive Associates (Other)
Responsible Party: Principal Investigator, Peter McGovern, MD, Medical Director, University Reproductive Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 0120100297
Record Dates: First submitted 2010-11-03; First posted 2010-11-09 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: PCOS; IVM; Polycystic ovarian syndrome; In Vitro Maturation; IVF
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- In Vitro Maturation (IVM) (Experimental)
  Interventions: Other: IVM

INTERVENTIONS:
Other: IVM — all patients in this pilot study will undergo IVM. IVM involves immature eggs being retrieved and matured in the laboratory.After maturation they are fertilized like is done in a typical IVF cycle.

SUMMARY:
This pilot study will be a prospective investigation to study the efficacy and safety of In-Vitro Maturation (IVM) for women with Polycystic Ovarian Syndrome (PCOS). There will be 10 subjects total in this Study. There will be no blinding to treatment.

In-Vitro Maturation will provide a viable, safe option for women with PCOS attempting pregnancy through the use of Assisted Reproductive Technology (ART).

ELIGIBILITY:
Inclusion Criteria

1. 10 women between the ages of 18-34 inclusive at time of signing Informed Consent Form.
2. A diagnosis of PCOS by their primary MD
3. An Antral Follicular Count (AFC) of > 12 on one ovary on at least one occasion
4. A day 3 FSH level of <8 IU/mL
5. In good general health off of current medications which may confound response to study medications.
6. Desire to seek pregnancy actively during the study period by IVF-ICSI.
7. A normal uterine cavity must have been confirmed by either hydrosonogram or hysteroscopy within two years of entering the study.
8. Male partner able to provide adequate semen sample by ejaculation (no TESE)

Exclusion Criteria

1. Current pregnancy
2. Patients with uncorrected thyroid disease (defined as TSH < 0.2 mIU/ML or >5.5 mIU/mL). A normal level within the last year is adequate for entry.
3. Patients with poorly controlled diabetes (HgB A1C over 8.0 ng/dL).
4. Patients enrolled simultaneously into other investigative studies that require medications, proscribe the study medications, limit intercourse, or otherwise prevent compliance with the protocol.
5. Patients with significant anemia (Hemoglobin < 10 mg/dL).
6. Patients enrolled simultaneously into other investigative studies that would interfere with this research study.
7. have any contraindications to using birth control pills (oral contraceptives) as determined by the attending physician (e.g. history of thromboembolism or estrogen-dependent malignancy, such as breast cancer, etc.) -

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Biochemical Pregnancy (defined as a rising Beta-HCG level). | 6 months

SECONDARY OUTCOMES:
number of immature oocytes retrieved | 6 months
rates of maturation and fertilization | 6 months
Incidence of Ovarian Hyperstimulation Syndrome (OHSS) | 6 months
live births | 1 1/2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. McGovern, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - University Reproductive Associates, Hasbrouck Heights, New Jersey
  - University Reproductive Associates, Hoboken, New Jersey